CLINICAL TRIAL: NCT01621503
Title: Prospective Comparative Clinical Study to Investigate the Use of the NON CONTACT TONO/PACHYMETER NT-530P
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nidek Co. LTD. (Industry)
Responsible Party: Sponsor
Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: NT530P-120210
Record Dates: First submitted 2012-06-14; First posted 2012-06-18 (Estimated); Last update posted 2013-06-28 (Estimated); Status verified 2012-07

CONDITIONS: IOP Ranges(mmHg): 7 to 16, >16 to <23, and 23 or More

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: NT-530P — intraocular pressure and central corneal thickness measurement

SUMMARY:
The primary objective of this clinical study is to collect clinical data to support an FDA 510(k) submission for the Nidek Non Contact Tono/ Pachymeter NT-530P. The secondary objective is to evaluate any adverse events found during the clinical study.

DETAILED DESCRIPTION:
Following data analysis will be conducted for tonometer and pachymeter readings. One of eyes of one patient becomes an object of the analysis. Regarding the intraocular pressure, higher IOP readings of either right or left eye are used for analysis. Regarding CCT, the readings of either right or left eye are randomly assigned to analysis in the order of registration.

ELIGIBILITY:
Inclusion Criteria:

1. IOP Measurement 1. 20 years or older who voluntarily agree to participate in this study after receiving adequate explanation 2. Possible to participate in the study regardless of existence of glaucoma
2. CCT Measurement 1. 20 years or older who voluntarily agree to participate in this study after receiving adequate explanation 2. Possible to participate in the study regardless of existence of glaucoma 3. Possible to participate in the study regardless of existence of corneal diseases (such as Keratoconus, post-LASIK, and corneal scars)

Exclusion Criteria:

1. IOP Measurement 1. Those with only one functional eye 2. Those with one eye having poor or eccentric fixation 3. Those with corneal scarring or who have had corneal surgery such as laser surgery 4. Microphthalmus 5. Buphthalmos 6. Contact lens wearers 7. Dry eyes 8. Blepharospasm 9. Nystagmus 10. Keratoconus 11. Those who have been diagnosed as having corneal conjunctivitis or other infectious disease 12. Those with central corneal thickness greater than 600 μm or less than 500 μm 13. A subject judged to be ineligible for participating in the study by the physicians in charge
2. CCT Measurement 1. Those with only one functional eye 2. Those with one eye having poor or eccentric fixation 3. Blepharospasm 4. Nystagmus 5. Those who have been diagnosed as having corneal conjunctivitis or other infectious disease 6. A subject judged to be ineligible for participating in the study by the physicians in charge

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2011-04; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
central corneal thickness | one day
intraocular pressure | one day

CONTACTS AND LOCATIONS:
Locations (2):
- Japan (2):
  - Kaiya ophthalmological clinic, Hamamatsu, Shizuoka
  - Ochanomizu Inoue ophthalmological clinic, Tokyo